CLINICAL TRIAL: NCT04834141
Title: Correlation Between Thoracic Kyphosis Posture and Static Balance
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2020.897
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Kyphosis; Balance; Distorted; Postural Kyphosis; Spine Disease; Balance
MeSH Terms: conditions — Kyphosis; Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kyphotic Group: Participants with kyphosis angle ≥ 40 degrees joined the kyphosis group. FlexiCurve ruler method was used, which is a reliable tool for measuring kyphosis height and kyphosis index. In addition, it is non-invasive, inexpensive, and easy to use in a clinical setting.
  Static balance Assessment:
  Objective evaluation of the static balance evaluated by the NeuroCom Balance Manager System ® static posturography device (45 × 45 cm NeuroCom® System Version 8.1 Balance Manager International, Clackamas, Oregon, USA)
  Interventions: Other: FlexiCurve ruler method to assess thoracic kyphosis angle
- Control Group: Participants with kyphosis angle < 40 degrees for the control group. FlexiCurve ruler method was used, which is a reliable tool for measuring kyphosis height and kyphosis index. In addition, it is non-invasive, inexpensive, and easy to use in a clinical setting.
  Static balance Assessment:
  Objective evaluation of the static balance evaluated by the NeuroCom Balance Manager System ® static posturography device (45 × 45 cm NeuroCom® System Version 8.1 Balance Manager International, Clackamas, Oregon, USA)
  Interventions: Other: FlexiCurve ruler method to assess thoracic kyphosis angle

INTERVENTIONS:
Other: FlexiCurve ruler method to assess thoracic kyphosis angle — The determination that the effect of thoracic kyphosis posture on trunk biomechanical alignment may be related to balance may contribute to new treatment recommendations in this area. The aim of this study is to investigate whether the thoracic kyphosis posture has an effect on static balance.
  Other Names: NeuroCom Balance Manager System ® static posturography device to assess static balance

SUMMARY:
The effects of balanced posture and postural changes have been evaluated in specific populations with different factors that can affect body postures and balance, such as age, musculoskeletal system, and other metabolic diseases. Studies on postural kyphosis and balance involvement are very few in the literature especially in the health population. Of the few studies that have evaluated kyphosis and balance, most are limited by small sample size and the exclusion of men. Many have focused primarily on the geriatric population. The determination that the effect of thoracic kyphosis posture on trunk biomechanical alignment may be related to balance may contribute to new treatment recommendations in this area. The aim of this study is to investigate whether the thoracic kyphosis posture has an effect on static balance.

DETAILED DESCRIPTION:
Background:

Kyphosis is roughly a slight forward curvature of the spine. A slight kyphosis or posterior curvature is normal throughout the human body and is present in every individual. Hyperkyphotic is a kyphotic angle greater than 40° commonly measured on a lateral X-ray measured by the Cobb method between C7 and T12. Postural stability or balance is the ability to keep the center of mass within the boundaries of the support base. Moving the center of mass beyond the boundaries of the support base may cause postural instability and loss of balance. There are studies showing that kyphotic posture affects the center of gravity and affects fall in the elderly, but there are limited studies on the effect of balance in young individuals.

The Aim of This Study Is:

To study the correlation between the balance and severity of thoracic kyphosis will be investigated

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over willing to attend the study.
* For those who join the thoracic kyphosis group, individuals with a kyphosis angle ≥ 40 degrees.
* Individuals with a kyphosis angle < 40 degrees for the control group.

Exclusion Criteria:

* Spine trauma, surgery, bone pathology, arthritis etc. have a history of illness Kyphotic deformity types are rounded back, Scheuermann's disease, hunched back, flat back and Dowager hump.
* Any spinal deformity, bone abnormality, postural deformity and disc herniation with / without peripheral symptoms.
* Body mass index (BMI), which is an indicator of obesity, is more than > 30.
* Complaining of balance problems, coordination problems, other neurological or vestibular diseases that affect body balance and posture.
* Having any orthopedic or neurological disease that affects the body joints or the integrity of the musculoskeletal system.
* Use of any medication that can cause dizziness or drowsiness in the last months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fourty-six subjects who joined the study were healthy without any disease might affect balance, body posture, and denied a past history of vestibular disorders, syncope, seizures, or neurological disorders such as stroke or Parkinson's disease.
  The study take place in Marmara university, Başıbüyük campus, between the period September 2020 to December 2020. Participants were recruited through online poster announcement, they directly contacted the primary investigator for booking an appointment. An appointment were made for the participants in the Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Biomechanics and Performance Analysis Laboratory, Marmara University.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Kyphosis Angle | 2 Months
  Kyphosis angle will be measured by felxicurve ruler, normally kyphosis angle below 40 degrees recognized as normal. For participants with kyphosis angle above 40 degrees recognized as hyperkyphotic posture. FlexiCurve ruler method is valid and reliable to the gold standard.
Static Balance Measures | 2 Months
  NeuroCom Balance Manager System ® static posturography device to assess static balance, which is objective evaluating system. The system compare the values reported for participants assessment then compare them to pre-recorded data base. The values of the test is assessed according to the percentage to the normal (average) values matched with the age group and gender. Above 80% determined as normal, and below this value determine balance disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: AYSEL yildiz, Ass. Prof., Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)